CLINICAL TRIAL: NCT05879536
Title: The Effect of Intravenous Infusion of Tramadol-ondansetron on Recovery After Caesarean Section. A Prospective, Observational and Non-inferiority Study Against Epidural Analgesia.
Brief Title: The Effect of Intravenous Infusion of Tramadol-ondansetron on Recovery After Caesarean Section.
Acronym: TRON
Status: Completed | Type: Observational
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Oscar Diaz-Cambronero, Principal Investigator. Head of the perioperative medicine group. Coordinator of the Clinical Medicine Unit, Hospital Universitario La Fe
Other Study IDs: TRON
Record Dates: First submitted 2023-04-04; First posted 2023-05-30 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Post Operative Pain; Cesarean Section; Tramadol; Postoperative Recovery; Quality of Recovery; Ondansetron; QoR-15; ObsQor-10; Postcesarean Recovery
Keywords: tramadol; cesarean section; postcesarean section; Qor-15; ObsQor-10; postcesarean recovery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- TRON (Tramadol-Ondansetron): Women who receive an infusion of tramadol-ondansetron from the end of the cesarean section and for the following 24 h. The infusion (TRON) is composed of 300 mg of tramadol and 12 mg of ondansetron dissolved in 250 ml of 0.9% saline, which is routinely programmed at 11 ml/h until the content is exhausted (approximately 23 hours).
  Interventions: Drug: Tramadol-ondansetron continuous infusion
- AL-EPI (Local anesthetics via epidural): Women who maintain the epidural catheter as the main measure of analgesia for 24 h. The epidural catheter after caesarean section is programmed with a 0.2% ropivacaine PCA (Patient controlled analgesia) pump at 7 ml/h with 7 ml on-demand boluses, with block every 20 min.
  Interventions: Drug: Ropivacaine via epidural catheter

INTERVENTIONS:
Drug: Tramadol-ondansetron continuous infusion — Analgesia strategy determined by routine use according to protocols, without investigator intervention.
  Groups: TRON (Tramadol-Ondansetron)
Drug: Ropivacaine via epidural catheter — Analgesia strategy determined by routine use according to protocols, without investigator intervention.
  Groups: AL-EPI (Local anesthetics via epidural)

SUMMARY:
It will be a prospective observational cohort study. The investigators will compare post-cesarean section recovery in patients receiving intravenous infusion of tramadol-ondansetron versus epidural catheter with infusion of local anesthetics.

DETAILED DESCRIPTION:
The primary outcome is to assess the non-inferiority in terms of post-cesarean section recovery of the intravenous perfusion of tramadol + ondansetron compared to the perfusion of local anesthetics through an epidural catheter.

This will be a prospective observational cohort study, with a total N of 312 patients who underwent a cesarean section. 156 who maintain the epidural catheter as the main measure of analgesia for 24 h, and 156 who receive an infusion of tramadol-ondansetron from the end of the cesarean section and for the following 24 h. The following data will be collected at 24 and 48 hours: need for unscheduled pharmacological reinforcement, adverse effects, QoR (Quality of Recovery) score 15, ObsQor-10 (Obstetric Quality of Recovery) score, and Visual Analogue Pain Scale (VAS) every 4 hours for 48 hours. The incidence of chronic pain 90 days after cesarean section will be assessed using the Numerical Pain Rating Scale (NRS).

ELIGIBILITY:
Inclusion Criteria:

* Woman over 18 years old undergoing caesarean section
* She agrees to participate voluntarily.
* She is already receiving any of the analgesic strategies studied.

Exclusion Criteria:

* Receiving an analgesic medication other than the one mentioned as "routine multimodal analgesia" (either as regular medication or for acute post-surgical pain)
* Medical history that determines the baseline data of the scales and data that we collect ( pain or previous disabilities; addiction to drugs, alcohol or drugs; another disease that worsens the quality of life)
* Medical history that conditions the pharmacological effect (allergy, intolerance or atypical reaction to any of the drugs involved in its treatment or possible cross-reactions )
* Contraindication for neuraxial techniques (patient refusal, difficulty in understanding or communication, localized infection, increased intracranial pressure, or other medical criteria)
* Two or more previous caesarean sections
* Difficulty in understanding or communication
* Mother care will not be available to the newborn in the postpartum period for any reason

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: The target population of this study would correspond to women who underwent a caesarean section (therefore, of childbearing age) in the first 48 hours of their puerperium, who underwent surgery at the HUiP La Fe. Among these, the patients who, following the practice usual clinical presentation in a standard cesarean section at the study center, receive a TRON or an infusion through the epidural catheter with ropivacaine.
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Post-surgical recovery | Day 1
  QoR-15 score at 24 hours after cesarean section

SECONDARY OUTCOMES:
Analgesia for acute pain | Day 1
  Pain score evolution on the sequential Visual Analogue Scale at 24 hours, measured every 4 hours.
Adverse effects | Day 1
  Presence or absence of the next adverse effects: Pruritus; tremors; urinary retention or need for a bladder catheter; Constipation or abdominal distension; limitation of mobility; delayed initiation of breastfeeding if desired (due to analgesia); need for blood extraction for control analysis.
Quality of recovery using ObsQoR10 - Spanish version | Day 1
  ObsQor-10 score at 24 hours.
Post-surgical recovery | Day 2
  QoR-15 score at 48 hours after cesarean section
Adverse effects | Day 2
  Presence or absence of the next adverse effects: Pruritus; tremors; urinary retention or need for a bladder catheter; Constipation or abdominal distension; limitation of mobility; delayed initiation of breastfeeding if desired (due to analgesia); need for blood extraction for control analysis.
Analgesia for acute pain | Day 2
  Pain score evolution on the sequential Visual Analogue Scale at 48 hours, measured every 4 hours.
Chronic Pain | Day 90
  Chronic pain measured by numerical rating scale at 90 days of TRON versus AL-EPI.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Myles PS, Boney O, Botti M, Cyna AM, Gan TJ, Jensen MP, Kehlet H, Kurz A, De Oliveira GS Jr, Peyton P, Sessler DI, Tramer MR, Wu CL; StEP-COMPAC Group; Myles P, Grocott M, Biccard B, Blazeby J, Boney O, Chan M, Diouf E, Fleisher L, Kalkman C, Kurz A, Moonesinghe R, Wijeysundera D. Systematic review and consensus definitions for the Standardised Endpoints in Perioperative Medicine (StEP) initiative: patient comfort. Br J Anaesth. 2018 Apr;120(4):705-711. doi: 10.1016/j.bja.2017.12.037. Epub 2018 Feb 2. PMID 29576111
- [Background] Moonesinghe SR, Jackson AIR, Boney O, Stevenson N, Chan MTV, Cook TM, Lane-Fall M, Kalkman C, Neuman MD, Nilsson U, Shulman M, Myles PS; Standardised Endpoints in Perioperative Medicine-Core Outcome Measures in Perioperative and Anaesthetic Care (StEP-COMPAC) Group. Systematic review and consensus definitions for the Standardised Endpoints in Perioperative Medicine initiative: patient-centred outcomes. Br J Anaesth. 2019 Nov;123(5):664-670. doi: 10.1016/j.bja.2019.07.020. Epub 2019 Sep 5. PMID 31493848
- [Background] Boney O, Moonesinghe SR, Myles PS, Grocott MPW; StEP-COMPAC group. Core Outcome Measures for Perioperative and Anaesthetic Care (COMPAC): a modified Delphi process to develop a core outcome set for trials in perioperative care and anaesthesia. Br J Anaesth. 2022 Jan;128(1):174-185. doi: 10.1016/j.bja.2021.09.027. Epub 2021 Nov 2. PMID 34740438
- [Background] Ma J, Martin R, Chan B, Gofeld M, Geary MP, Laffey JG, Abdallah FW. Using Activity Trackers to Quantify Postpartum Ambulation: A Prospective Observational Study of Ambulation after Regional Anesthesia and Analgesia Interventions. Anesthesiology. 2018 Mar;128(3):598-608. doi: 10.1097/ALN.0000000000001979. PMID 29135475
- [Background] Delfino E, Netto R, Zanon D. Pain control after cesarean delivery: a new proposal for a continuous locoregional technique. Int J Obstet Anesth. 2021 Nov;48:103196. doi: 10.1016/j.ijoa.2021.103196. Epub 2021 Jun 23. No abstract available. PMID 34243070
- [Background] Practice Guidelines for Obstetric Anesthesia: An Updated Report by the American Society of Anesthesiologists Task Force on Obstetric Anesthesia and the Society for Obstetric Anesthesia and Perinatology. Anesthesiology. 2016 Feb;124(2):270-300. doi: 10.1097/ALN.0000000000000935. No abstract available. PMID 26580836
- [Background] Vercauteren M, Vereecken K, La Malfa M, Coppejans H, Adriaensen H. Cost-effectiveness of analgesia after Caesarean section. A comparison of intrathecal morphine and epidural PCA. Acta Anaesthesiol Scand. 2002 Jan;46(1):85-9. doi: 10.1034/j.1399-6576.2002.460115.x. PMID 11903078
- [Background] Chi X, Li M, Mei W, Liao M. Comparison of patient-controlled intravenous analgesia with sufentanil versus tramadol in post-cesarean section pain management and lactation after general anesthesia - a prospective, randomized, double-blind, controlled study. J Pain Res. 2017 Jul 3;10:1521-1527. doi: 10.2147/JPR.S137799. eCollection 2017. PMID 28740418
- [Background] Duan G, Bao X, Yang G, Peng J, Wu Z, Zhao P, Zuo Z, Li H. Patient-controlled intravenous tramadol versus patient-controlled intravenous hydromorphone for analgesia after secondary cesarean delivery: a randomized controlled trial to compare analgesic, anti-anxiety and anti-depression effects. J Pain Res. 2018 Dec 18;12:49-59. doi: 10.2147/JPR.S184782. eCollection 2019. PMID 30588079
- [Background] Siddik-Sayyid S, Aouad-Maroun M, Sleiman D, Sfeir M, Baraka A. Epidural tramadol for postoperative pain after Cesarean section. Can J Anaesth. 1999 Aug;46(8):731-5. doi: 10.1007/BF03013907. PMID 10451131
- [Background] Nnacheta TE, Onyekwulu FA, Amucheazi AO. Prevention of postanesthetic shivering under subarachnoid block for cesarean section: A randomized, controlled study comparing tramadol versus ondansetron. Niger J Clin Pract. 2020 May;23(5):619-625. doi: 10.4103/njcp.njcp_641_18. PMID 32367867
- [Background] Jayaraj A, Balachander H, Kuppusamy SK, Arusamy S, Rai Y, Siddiqui N. Comparison of meperidine, tramadol and fentanyl for post-spinal shivering prevention during cesarean delivery: A double-blind randomized controlled trial. J Obstet Gynaecol Res. 2019 Nov;45(11):2202-2208. doi: 10.1111/jog.14106. Epub 2019 Sep 4. PMID 31486253
- [Background] Sammour RN, Ohel G, Cohen M, Gonen R. Oral naproxen versus oral tramadol for analgesia after cesarean delivery. Int J Gynaecol Obstet. 2011 May;113(2):144-7. doi: 10.1016/j.ijgo.2010.11.024. PMID 21435642
- [Background] Sahmeddini MA, Azemati S, Motlagh EM. Local Infiltration of Tramadol versus Bupivacaine for Post Cesarean Section Pain Control: A Double-Blind Randomized Study. Iran J Med Sci. 2017 May;42(3):235-241. PMID 28533571
- [Background] Mitra S, Khandelwal P, Sehgal A. Diclofenac-tramadol vs. diclofenac-acetaminophen combinations for pain relief after caesarean section. Acta Anaesthesiol Scand. 2012 Jul;56(6):706-11. doi: 10.1111/j.1399-6576.2012.02663.x. Epub 2012 Mar 5. PMID 22385415
- [Background] Wu Z, Zhao P, Peng J, Fang L, Ding J, Yan G, Wang Y, Zhu J, Wang D, Li Y, Chen Z, Zhang Q, Deng Q, Duan G, Zuo Z, Li H. A Patient-Controlled Intravenous Analgesia With Tramadol Ameliorates Postpartum Depression in High-Risk Woman After Cesarean Section: A Randomized Controlled Trial. Front Med (Lausanne). 2021 May 27;8:679159. doi: 10.3389/fmed.2021.679159. eCollection 2021. PMID 34124111
- [Background] Weibel S, Neubert K, Jelting Y, Meissner W, Wockel A, Roewer N, Kranke P. Incidence and severity of chronic pain after caesarean section: A systematic review with meta-analysis. Eur J Anaesthesiol. 2016 Nov;33(11):853-865. doi: 10.1097/EJA.0000000000000535. PMID 27635953
- [Background] Johansen A, Schirmer H, Nielsen CS, Stubhaug A. Persistent post-surgical pain and signs of nerve injury: the Tromso Study. Acta Anaesthesiol Scand. 2016 Mar;60(3):380-92. doi: 10.1111/aas.12653. Epub 2015 Nov 5. PMID 26537886
- [Background] Richez B, Ouchchane L, Guttmann A, Mirault F, Bonnin M, Noudem Y, Cognet V, Dalmas AF, Brisebrat L, Andant N, Soule-Sonneville S, Dubray C, Duale C, Schoeffler P. The Role of Psychological Factors in Persistent Pain After Cesarean Delivery. J Pain. 2015 Nov;16(11):1136-46. doi: 10.1016/j.jpain.2015.08.001. Epub 2015 Aug 20. PMID 26299436
- [Background] Borges NC, de Deus JM, Guimaraes RA, Conde DM, Bachion MM, de Moura LA, Pereira LV. The incidence of chronic pain following Cesarean section and associated risk factors: A cohort of women followed up for three months. PLoS One. 2020 Sep 4;15(9):e0238634. doi: 10.1371/journal.pone.0238634. eCollection 2020. PMID 32886704
- [Background] Lavand'homme P. Postpartum chronic pain. Minerva Anestesiol. 2019 Mar;85(3):320-324. doi: 10.23736/S0375-9393.18.13060-4. Epub 2018 Oct 30. PMID 30394066
- [Background] Morales-Ariza V, Loaiza-Aldean Y, de Miguel M, Pena-Navarro M, Martinez-Silva O, Gonzalez-Tallada A, Manrique-Munoz S, de Nadal M. Validation and cross-cultural adaptation of the postoperative quality of recovery 15 (QoR-15) questionnaire for Spanish-speaking patients: A prospective cohort study. Am J Surg. 2023 Apr;225(4):740-747. doi: 10.1016/j.amjsurg.2022.11.009. Epub 2022 Nov 17. PMID 36414472
- [Background] Ciechanowicz S, Setty T, Robson E, Sathasivam C, Chazapis M, Dick J, Carvalho B, Sultan P. Development and evaluation of an obstetric quality-of-recovery score (ObsQoR-11) after elective Caesarean delivery. Br J Anaesth. 2019 Jan;122(1):69-78. doi: 10.1016/j.bja.2018.06.011. Epub 2018 Jul 31. PMID 30579408
- [Background] Ciechanowicz S, Howle R, Heppolette C, Nakhjavani B, Carvalho B, Sultan P. Evaluation of the Obstetric Quality-of-Recovery score (ObsQoR-11) following non-elective caesarean delivery. Int J Obstet Anesth. 2019 Aug;39:51-59. doi: 10.1016/j.ijoa.2019.01.010. Epub 2019 Feb 2. PMID 30885691
- [Background] Sultan P, Kamath N, Carvalho B, Bansal P, Elkhateb R, Dougan S, Whittington J, Guo N, El-Sayed Y, Mhyre J, Sharawi N. Evaluation of inpatient postpartum recovery using the Obstetric Quality of Recovery-10 patient-reported outcome measure: a single-center observational study. Am J Obstet Gynecol MFM. 2020 Nov;2(4):100202. doi: 10.1016/j.ajogmf.2020.100202. Epub 2020 Aug 17. PMID 33345919
- [Background] Sultan P, Kormendy F, Nishimura S, Carvalho B, Guo N, Papageorgiou C. Comparison of spontaneous versus operative vaginal delivery using Obstetric Quality of Recovery-10 (ObsQoR-10): An observational cohort study. J Clin Anesth. 2020 Aug;63:109781. doi: 10.1016/j.jclinane.2020.109781. Epub 2020 Mar 20. PMID 32203873
- [Background] Mathias LAST, Carlos RV, Siaulys MM, Gabriades P, Guo N, Domingue B, O'Carroll J, Carvalho B, Sultan P. Development and validation of a Portuguese version of Obstetric Quality of Recovery-10 (ObsQoR-10-Portuguese). Anaesth Crit Care Pain Med. 2022 Jun;41(3):101085. doi: 10.1016/j.accpm.2022.101085. Epub 2022 Apr 26. PMID 35487408
- [Background] Kozanhan B, Yildiz M, Polat A, Gunenc O, Tutar SM, Iyisoy MS, Kulhan NG, Sultan P. Development and Validation of a Turkish Version of Obstetric Quality of Recovery-10. Turk J Anaesthesiol Reanim. 2022 Oct;50(5):366-372. doi: 10.5152/TJAR.2022.21441. PMID 36301286

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-08-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT05879536/SAP_000.pdf